CLINICAL TRIAL: NCT04032964
Title: A Dose Finding Study of the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF in Combination With Doxorubicin in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Dose Finding Study of L19TNF and Doxorubicin in Patients With STS
Acronym: DOXO75
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFDOX75-02/19
Record Dates: First submitted 2019-06-28; First posted 2019-07-25 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Intervention Model Description: Open-label, phase 1 dose confirmation study in patients with advanced, unresectable and/or metastatic soft tissue sarcoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm L19TNF + DOXO (Experimental): Patients will be treated with:
  * doxorubicin 75 mg/m2 i.v. on day 1 of each 21-day cycle;
  * L19TNF 13 µg/kg i.v. on day 1, 3 and 5 of each 21-day cycle
  Interventions: Drug: L19TNF; Drug: DOXORUBICIN

INTERVENTIONS:
Drug: L19TNF — L19TNF 13 µg/kg i.v. will be administered on day 1, 3 and 5 of each 21-day cycle
Drug: DOXORUBICIN — Doxorubicin 75 mg/m2 will be administered on day 1 of each 21-day cycle

SUMMARY:
The study is aimed at evaluating the safety of L19TNF in combination with the most appropriate dose of doxorubicin.

DETAILED DESCRIPTION:
Open-label, phase 1 dose confirmation study in patients with advanced, unresectable and/or metastatic soft tissue sarcoma.

Six (6) Patients will be enrolled sequentially and will be treated according to the following scheme:

• Doxorubicin 75 mg/m2 i.v. on day 1 of each 21-day cycle L19TNF 13 µg/kg i.v. on day 1,3 and 5 of each 21-day cycle Initiation of the study treatment for an individual subject will occur no less than 3 days after initiation of the study treatment for the previous patient. Not more than 2 patients are to be treated simultaneously in Cycle 1.

Should unacceptable toxicities occur in ≥ 2 patients during the observation period from Day 1 to Day 21 (first cycle), enrollment will be stopped.

If a patient is not evaluable for unacceptable toxicity, he/she will be replaced.

Patients will be treated in repeated cycles until the treatment or when one of the following criteria are met:

* Unacceptable toxicity
* Disease Progression or relapse
* The patient or the investigator requests the treatment discontinuation
* The patient meets a withdrawal criterion. Patients with SD or PR (according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 evaluation) after the maximum of 6 cycles of study treatment, will receive maintenance therapy for up to 18 maintenance cycles from start of treatment, toxicity or until disease progression occurs. Maintenance can start immediately after the end of cycle 6 and consists infusions of L19TNF on Day 1 of each maintenance cycle (every 3 weeks) and doxorubicin on Day 1 of maintenance cycle 1 and 2 (if appropriate).

The primary objective is to evaluate the safety of L19TNF in combination with doxorubicin and to establish a recommended dose (RD), assessed as follows:

* Adverse events (AEs), serious adverse events (SAE) and drug induced liver injury (DILI) assessment based on Common Terminology Criteria for Adverse Events (CTCAE) v.5.0
* Standard laboratory (hematology, biochemistry and urinalysis) parameters.
* Electrocardiogram (ECG) and echocardiogram (ECHO) findings. In particular, data about QT/QTc intervals will be collected and analyzed for QT/QTc prolongation potentially caused by treatment.
* Physical examination findings including assessment of vital signs and physical measurements.

The secondary objective of the study is to evaluate signs of efficacy measured as progression-free survival (PFS) rate at 3, 6, 9, 12 and 18 months.

The other secondary objectives of the study are as follows:

* Efficacy of L19TNF in combination with doxorubicin:
* Overall response rate (ORR, consisting of CR and PR).
* Disease Control Rate (DCR, i.e. complete response (CR), partial response (PR) and stable disease (SD))
* Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19TNF.
* Characterization of pharmacokinetics (PK) of L19TNF and doxorubicin

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years.
2. Histologically confirmed diagnosis of advanced unresectable or metastatic soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy. Participants with Kaposi's sarcoma and gastrointestinal stromal tumors (GIST) will be excluded. Note: Evidence of disease progression is required for participants that are not newly diagnosed.
3. Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria 1.1. If only one lesion is present at screening this lesion should not have been irradiated during previous treatments.
4. Life expectancy of at least 3 months in the judgment of the investigator.
5. ECOG ≤ 2.
6. Documented negative test for HIV-HBV-HCV. For HBV serology: the determination of HBsAg, anti-HBsAg-Ab and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
7. Female patients: negative serum pregnancy test for women of childbearing potential (WOCBP)* within 14 days of starting treatment. WOCBP must agree to use, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence. Male patients: Male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required.
8. Informed consent signed and dated to participate in the study.
9. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

   * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)

Exclusion Criteria:

1. Diagnosis of GIST or Kaposi sarcoma.
2. Prior therapy (except surgery and radiation) for this presentation of unresectable or metastatic malignant soft tissue sarcoma.
3. Previous treatment with anthracycline- or anthracenedione-containing chemotherapy.
4. Radiotherapy within 3 weeks (21 days) prior to therapy and previous radiation therapy to the mediastinal or pericardial area.
5. Active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis). Participants with a history of a CNS metastasis previously treated with curative intent (for example, stereotactic radiation or surgery) that have not progressed on follow-up imaging, have been asymptomatic for at least 60 days and are not receiving systemic corticosteroids and or/anticonvulsants, are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before randomization to rule out brain metastasis.
6. Known history of allergy to TNF, anthracyclines, or other intravenously administered human proteins/peptides/antibodies.
7. Absolute neutrophil count (ANC) < 1.5 x 109/L, platelets < 100 x 109/L and hemoglobin (Hb) < 9.0 g/dl.
8. Chronically impaired renal function as expressed by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
9. Inadequate liver function (ALT, AST, ALP or total bilirubin ≥ 2.5 x ULN).
10. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
11. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
12. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
13. Clinically significant cardiac arrhythmias or requiring permanent medication.
14. Abnormalities observed during baseline ECG and ECHO investigations that are considered as clinically significant by the investigator. Subjects with current, or a history of QT/QTc prolongation would be excluded. In particular:

    * patients with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of QTc >480 milliseconds using Fredricia's QT correction formula) are excluded;
    * patients with a history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of prolonged QT syndrome) are excluded;
    * patients who require the use of concomitant medications that prolong the QT/QTc interval are excluded.
15. Uncontrolled hypertension.
16. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
17. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
18. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
19. Pregnancy or breast-feeding.
20. Requirement of chronic administration of corticosteroids or other immunosuppressant drugs. Limited use of corticosteroids to treat or prevent infusion-related reactions and hypersensitivity reactions is not considered an exclusion criterion.
21. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
22. Known active or latent tuberculosis (TB).
23. Concurrent malignancies other than soft tissue sarcoma, unless the patient has been disease-free for at least 2 years.
24. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
25. Serious, non-healing wound, ulcer or bone fracture.
26. Allergy to study medication or excipients in study medication.
27. Concurrent therapy with anticoagulants.
28. Concurrent use of other anti-cancer treatments or agents other than study medication.
29. Any recent live vaccination within 4 weeks prior to treatment or plan to receive vaccination during the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number and type of Adverse events (AE) | From week 1 to week 72
  Adverse event (AE) for the assessment of safety (CTCAE v. 5.0)
Number and type of Serious Adverse events (SAE) | From week 1 to week 72
  Serious Adverse Events (SAE) for the assessment of safety (CTCAE v. 5.0)
Number and type of Drug induced liver injury (DILI) | From week 1 to week 72
  Drug induced liver injury (DILI) assessment based on CTCAE v.5.0
Electrocardiogram (ECG) findings | From week 1 to week 72
  Electrocardiogram (ECG) findings. In particular, data about QT/QTc intervals will be collected and analyzed for QT/QTc prolongation potentially caused by treatment.
Echocardiogram (ECHO) findings | From week 1 to week 72
  Echocardiogram (ECHO) findings. In particular, data about QT/QTc intervals will be collected and analyzed for QT/QTc prolongation potentially caused by treatment.
Calculation of the body surface area (BSA) | From week 1 to week 72
  BSA
Measurement of body weight | From week 1 to week 72
  Measurement of body weight
Heart rate | From week 1 to week 72
  Measurement of heart rate
Blood pressure | From week 1 to week 72
  Measurement of blood pressure
ECOG performance status | From week 1 to week 72

SECONDARY OUTCOMES:
Progression-free survival (PFS) rate | 3, 6, 9, 12 and 18 months
  To evaluate signs of efficacy measured as progression-free survival (PFS) rate
Efficacy of L19TNF in combination with doxorubicin: Overall response rate | 3, 6, 9, 12 and 18 months
  Overall response rate (ORR, consisting of CR and PR)
Efficacy of L19TNF in combination with doxorubicin: Disease Control Rate | 3, 6, 9, 12 and 18 months
  Disease Control Rate (DCR, consisting of CR, PR and SD)
HAFA measurement | Treatment phase: at day 1 of cycle 1, at day 8 of week 1, at day 1 of cycle 2 and at day 1 of every cycle; at day 1 of every maintenance cycle (each cycle is 21 days)
  Assessment of the formation of Human anti-fusion protein antibodies (HAFA) against L19TNF
PK value of L19TNF | Cycle 1 day 1, Cycle 1 day 2, cycle 1 day 3 and cycle 1 day 5 (each cycle is 21 days)
  Measurement of AUC value of L19TNF
PK value of doxorubicin | Cycle 1 day 1, Cycle 1 day 2, cycle 1 day 3 and cycle 1 day 5 (each cycle is 21 days)
  Measurement of AUC value of doxorubicin

CONTACTS AND LOCATIONS:
Locations (1):
- Sarcoma Oncology Research Center (SORC) Cancer Center of Southern California, Santa Monica, California, United States